CLINICAL TRIAL: NCT00300846
Title: A Multicenter, Comparative, Randomized, Double-Blind, Placebo Controlled Study on the Effect on Weight of Adjunctive Treatment With Aripiprazole in Patients With Schizophrenia.
Brief Title: A Study of Adjunctive Treatment of Aripiprazole in Schizophrenic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN138-170
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2008-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A1 (Active Comparator)
  Interventions: Drug: aripiprazole
- A2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: aripiprazole — Tablets, Oral, 5 mg, 10 mg, 15 mg, once daily, 16 weeks followed by 12 weeks of Open-Label extension phase (optional).
  Other Names: Abilify
  Arms: A1
Drug: Placebo — Tablets, Oral, 0 mg, once daily, 16 weeks followed by 12 weeks of Open-Label extension phase (optional)
  Arms: A2

SUMMARY:
The purpose of this study is to evaluate the effect on patient weight of adjunctive therapy of aripiprazole with clozapine versus clozapine monotherapy, in schizophrenic patients who are not optimally controlled on clozapine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia treated with clozapine (200-900 mg/day), who gained at least 2.5 kg while on clozapine.

Exclusion Criteria:

* Patients known to be allergic to aripiprazole
* Hospitalized patients
* Patients who have previously received study medication in an aripiprazole clinical study or who have participated in any clinical trial with an investigational agent within the past month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Evaluate effect on patient weight of adjunctive therapy of aripiprazole with clozapine versus clozapine mono-therapy in schizophrenic patients who are not optimally controlled on clozapine.
The mean change from baseline in patient weight at Week 16 (LOCF) will be compared between the 2 groups.

SECONDARY OUTCOMES:
Efficacy (PANSS, CGI)
Effectiveness (IAQ, GAF)
Patient Reported Outcomes
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (57):
- Austria (3):
  - Local Institution, Graz
  - Local Institution, Innsbruck
  - Local Institution, Vienna
- Czechia (5):
  - Local Institution, Brno-Bohunice
  - Local Institution, Hradec Králové
  - Local Institution, Litoměřice
  - Local Institution, Opava
  - Local Institution, Prague
- Finland (3):
  - Local Institution, Helsingin Kaupunki
  - Local Institution, Tampere
  - Local Institution, Turku
- France (9):
  - Local Institution, Brumath
  - Local Institution, Bully-les-Mines
  - Local Institution, Clermont-Ferrand
  - Local Institution, Limoges
  - Local Institution, Lyon
  - Local Institution, Nîmes
  - Local Institution, Paris
  - Local Institution, Rennex Cedex 7
  - Local Institution, Sotteville-lès-Rouen
- Germany (6):
  - Local Institution, Augsburg
  - Local Institution, Berlin
  - Local Institution, Duisburg
  - Local Institution, Haar
  - Local Institution, Heidelberg
  - Local Institution, Mannheim
- Hungary (2):
  - Local Institution, Budapest
  - Local Institution, Szolnok
- Poland (5):
  - Local Institution, Krakow
  - Local Institution, Leszno
  - Local Institution, Skorzewo
  - Local Institution, Torun
  - Local Institution, Warsaw
- South Africa (5):
  - Local Institution, Soweto, Gauteng
  - Local Institution, Vereeniging, Gauteng
  - Local Institution, Durban, KwaZulu-Natal
  - Local Institution, Bellville, Western Cape
  - Local Institution, Cape Town, Western Cape
- Sweden (9):
  - Local Institution, Bromma
  - Local Institution, Falköping
  - Local Institution, Linköping
  - Local Institution, Luleå
  - Local Institution, Malmo
  - Local Institution, Solna
  - Local Institution, Uppsala
  - Local Institution, Varberg
  - Local Institution, Västra Frölunda
- Local Institution, Bern, Switzerland
- Turkey (Türkiye) (3):
  - Local Institution, Antalya
  - Local Institution, Istanbul
  - Local Institution, Izmir
- United Kingdom (6):
  - Local Institution, Exeter, Devon
  - Local Institution, Teignmouth, Devon
  - Local Institution, Welwyn Garden City, Hertfordshire
  - Local Institution, Hull, North Yorkshire
  - Local Institution, Dundee, Tayside
  - Local Institution, London

REFERENCES:
- [Derived] Fleischhacker WW, Heikkinen ME, Olie JP, Landsberg W, Dewaele P, McQuade RD, Loze JY, Hennicken D, Kerselaers W. Effects of adjunctive treatment with aripiprazole on body weight and clinical efficacy in schizophrenia patients treated with clozapine: a randomized, double-blind, placebo-controlled trial. Int J Neuropsychopharmacol. 2010 Sep;13(8):1115-25. doi: 10.1017/S1461145710000490. Epub 2010 May 12. PMID 20459883